CLINICAL TRIAL: NCT00186134
Title: Walk to School and Physical Activity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 95378
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Physical Activity
Keywords: Physical Activity; Walking; Primary Schools; Transportation
MeSH Terms: conditions — Motor Activity | interventions — Exercise

INTERVENTIONS:
Behavioral: physical activity

SUMMARY:
The purpose of the proposed study is to determine the effect of walking to school for one week on total physical activity and patterns of physical activity in third, fourth and fifth grade students.

DETAILED DESCRIPTION:
Increasing children's physical activity has become an important public health concern. Active transportation (walking and bicycling) is one aspect of children's physical activity that has received little attention but may provide a means of increasing children's activity levels. Traveling to school is a common activity for most children in the United States. Due to this regularity, active transportation to school provides a possible way to incorporate an increase in children's moderate-to-vigorous physical activity into a routine activity.

Several "walk to school" programs have been implemented but it is not known if the physical activity levels of children walking to school are greater than those that get chauffeured or bused. Theoretically, moderate intensity activity should be greater in the walkers compared to others. This difference should be in proportion to the duration of the walk to and from school; determined by how far the child lives from the school. However, more activity in the morning may have an impact on activity levels later in the day. Therefore, differences in daily activity patterns in addition to total activity need to be considered.

Comparison(s): Following a baseline week, the physical activity of students randomized to a Walk to School group will be compared to those randomized to a Control group, who will continue to be driven to school.

ELIGIBILITY:
Inclusion Criteria:

* 3rd, 4th, or 5th grade at participating school

Exclusion Criteria:

* Currently walking or bicycling to school at least 4 times per week
* Physical or mental disability that would prevent walking to school under adult supervision.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30
Dates: Start 2004-10; Study Completion 2005-05

PRIMARY OUTCOMES:
Accelerometer derived average minutes of moderate-to-vigorous physical activity per day.
Accelerometer derived average counts per minute per day.

SECONDARY OUTCOMES:
Accelerometer derived average minutes of moderate-to-vigorous physical activity before, during, and after school and in the evening.
Accelerometer derived average counts per minute per day before, during, and after school and in the evening.

CONTACTS AND LOCATIONS:
Overall Officials: John R Sirard, PhD, Principal Investigator — Stanford University; Thomas N Robinson, MD, MPH, Study Director — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Boarnet MG, Anderson CL, Day K, McMillan T, Alfonzo M. Evaluation of the California Safe Routes to School legislation: urban form changes and children's active transportation to school. Am J Prev Med. 2005 Feb;28(2 Suppl 2):134-40. doi: 10.1016/j.amepre.2004.10.026. PMID 15694521
- [Background] Gordon-Larsen P, Nelson MC, Beam K. Associations among active transportation, physical activity, and weight status in young adults. Obes Res. 2005 May;13(5):868-75. doi: 10.1038/oby.2005.100. PMID 15919840
- [Background] Sirard JR, Ainsworth BE, McIver KL, Pate RR. Prevalence of active commuting at urban and suburban elementary schools in Columbia, SC. Am J Public Health. 2005 Feb;95(2):236-7. doi: 10.2105/AJPH.2003.034355. PMID 15671456